CLINICAL TRIAL: NCT00481260
Title: Characteristics of Hgb C Carriers in Northern Israel and Clinical Features Among Hgb Homozygous
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr Koren Ariel, Pediatric Hematology Unit - HaEmek Medical Center - Afula - Israel
Other Study IDs: 5100706.EMC
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Hgb C Hemoglobinopathy
Keywords: Hgb C; Screening
MeSH Terms: interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Medical history and basic laboratory analysis — Medical history and basic laboratory analysis

SUMMARY:
Hgb C is an hemoglobinopathy quite rare in Israel. The clinical status of patients that are diagnosed as homozygous to this disease is quite benign but not study in large groups.

Also the characteristics of carriers and the incidence in northern Israel were a large arab population lives, was not study. The results of this study can be useful for screening purpose in a area were another hemoglobinopathies are frequent.

DETAILED DESCRIPTION:
Hgb C is an hemoglobinopathy quite rare in Israel. The clinical status of patients that are diagnosed as homozygous to this disease is quite benign but not study in large groups.

Also the characteristics of carriers and the incidence in northern Israel were a large arab population lives, was not study. The results of this study can be useful for screening purpose in a area were another hemoglobinopathies are frequent.

The study will record the clinical characteristics of the homozygous Hgb C patients and the hematology characteristics of all the heterozygous carriers detected in northern Israel

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as homozygous for Hgb C disease or double heterozygous in combination to other abnormal hemoglobin, and all the carriers detected in the hematology laboratory during the screening for abnormal hemoglobins in northern Israel

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed at the pediatric Hematology Unit of laboratory data from the thalassemia screening in northern Israel
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; luci Zalman, Phd, Study Chair — Hematology Laboratory - HaeEmek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel